CLINICAL TRIAL: NCT05111756
Title: Braining Study - Implementation of Physical Activity for Patients and Staff in Specialist Psychiatry, Feasibility on Pilot Unit and Effect Evaluation in Randomized Controlled Multi-center Study.
Brief Title: Braining - Physical Exercise in Psychiatry - Evaluation of Feasibility, Implementation and Health Among Staff
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: Braining - personell
Record Dates: First submitted 2021-10-22; First posted 2021-11-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Physical Inactivity; Occupational Stress
Keywords: physical exercise; psychiatric staff; Occupational Stress; implementation; feasibility
MeSH Terms: conditions — Sedentary Behavior; Occupational Stress; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Unit A: Staff at first phase units, receiving Braining, physical exercise
- Unit B: Staff at second phase units, receiving Braining, physical exercise

SUMMARY:
Physical exercise (PE) shows beneficial effects on somatic and psychiatric symptoms. "Braining" is a clinical invention where psychiatric staff exercise together with patients to help patients start and execute PE regularly. In the present study feasibility of the intervention will be evaluated, how Braining is perceived and implemented, and effects on health and physical activity among staff. It is hypothesized that staff health and physical activity will increase after implementing Braining at the unit. Braining will be implemented at four psychiatric units in Region Stockholm, Sweden. During 6 months staff will be trained and receive implementation support. To measure feasibility the staff will answer self-rating questionnaires and be invited to a focus group interview post the implementation period. Implementation will be evaluated by ratings of compliance, the self-rating questionnaire Normalization Process Theory Measure (S-NoMAD), and focus group interviews. Health will be measured by self ratings of stress, sleep, general health, and engagement pre implementation and every month during the 6 month implementation phase. Ratings will be repeated at follow up 12 month after implementation started. Physical activity will be rated during the 6 months implementation phase using a tracker of activity and at follow up 12 month after implementation started. All staff at the units will be invited to participate in the evaluations, approximately 20 individuals per unit.

DETAILED DESCRIPTION:
"Braining" is a clinical invention that helps patients in psychiatry to start and execute physical exercise (PE) regularly in psychiatric care. The core components are basic high performance group training session and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care and is included in the patient care plan. Braining is unique in that it:

1. Includes trained psychiatric clinical staff exercising together with patients from both out- and inpatient ward units in daily, high endurance group training sessions
2. is included in regular healthcare fee, (free of charge)
3. includes a motivational and educational visit (as a group seminar or as an individual visit) at the start and end of a twelve week training period
4. includes regular measurements (self-assessment questionnaires, blood samples, physical and mental health examination and education before and after the twelve week training period)
5. offers short individual motivating visits before every training session, including assessment of day shape and fitness to participate.

In the present study focus is on the feasibility of the intervention, how Braining is perceived and implemented, and effects on health and physical activity among staff. The research questions are:

* How do staff experience Braining regarding acceptability, applicability and suitability?
* Is there a correlation between the staff's work with Braining and occupational health, measured as performed PE, perceived stress, and general health?
* Is there a correlation between the staff's work with Braining and occupational health, measured as exhaustion, sleep, sick leave, and job engagement?
* Is there a significant interaction effect between change over time in occupational health, measured with PSS-10 and GHQ, and participation in Braining sessions according to "Ratings of Braining sessions"?
* Is there a significant interaction effect between change over time on physical activity measured with Actigraph and IPAQ and participation in Braining sessions according to "Ratings of Braining sessions"?
* Is there an interaction effect between physical activity measured with Actigraph and IPAQ and occupational health measured with PSS-10 and GHQ?
* Does Braining have a specific effect for staff who during baseline rate over cut-off on GHQ and PSS-10 respectively?
* How compliant are staff to the Braining method in the sense of number completed training sessions, quality of completed sessions, compliance with the core components of the method?
* To what extent is Braining integrated into ordinary work at the unit in short (6 months) and long term (1 and 2 years)?

Braining is to be implemented at 4 psychiatric care units the upcoming years starting nov 2021. Approximately 20 personnel on each unit will be included. Planned design is a longitudinal pre-post study with four measurements during ongoing intervention (weeks 1, 4, 8 and 12) and two follow-ups (6 months and 12 months post inclusion). Improved design with three baseline observation (data points) and possible interrupted time series design, (ITSD). Relationships between the staff's work with Braining and their own occupational health are examined self-estimates, see list. Physical activity level is measured with activity tracker before training and measured throughout the 6 months and at follow-up after 12 months.

Experience of the implementation process is evaluated with S-NoMAD, which is administered at two occasions during the intervention, after completion and at follow-up after 2 years. Staff experience of working with Braining is examined with self-assessments and in focus group interviews after the end of the intervention. Staff compliance with Braining is evaluated based on a checklist where data is collected through weekly follow-ups of the work on the unit as well as observation of completed training sessions.

Data analysis Qualitative analysis: Recorded material from focus group interviews is transcribed and analyzed based on the thematic analysis method according to Braun & Clarke et al 2006). The method aims to understand the individual's perspective in relation to a particular phenomenon and is often used as an inductive hypothesis-generating approach.

Continuous data will be analyzed using mixed effects models or t-test, nominal data analyzed mainly with chi2 test. In mixed effects models of differences between groups the interaction effect of group and time will be the central estimate.

ELIGIBILITY:
Inclusion Criteria:

* Works at one of the relevant units regardless of occupational category, including administrative services.
* Permanent employment or fixed-term employment for at least one more year after the start of studies.

Exclusion Criteria:

* Medical conditions such as heart or lung disease, infection, abstinence where heart rate-increasing physical activity is considered contraindicated due to Medical reasons.
* Full-time sick leave> 1 month during the training period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Staff of a psychiatric care unit
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Minutes spent on Physical movement (high, moderate, low) | Change from baseline to follow up observation 6 months after inclusion
  Physical exercise conducted by staff, measured by actigraph
Minutes spent on Physical movement self rated (high, moderate, low) | Change from baseline to follow up observation 6 months after inclusion
  Physical exercise conducted by staff, measured by self ratings of International Physical Activity Questionnaires (IPAQ)
General health | Change from baseline to follow up observation 6 months after inclusion
  General health measured by self ratings of General health questionnaire (GHQ), scores 0-12, higher scores indicates more mental distress
Perceived stress | Change from baseline to follow up observation 6 months after inclusion
  Perceived stress measured by self ratings of Perceived stress scale (PSS-10), , scores 0-40, higher scores indicates more mental distress
Perceived feasibility of Intervention | 1 month after implementation start
  Feasibility measured by self ratings of Feasibility of Intervention Measure (FIM)
Perceived feasibility of Intervention | 6 months after implementation start
  Feasibility measured by self ratings of Feasibility of Intervention Measure (FIM)
Acceptability of Intervention | 1 month after implementation start
  Acceptability measured by self ratings of Acceptability of Intervention Measure (AIM)
Acceptability of Intervention | 6 months after implementation start
  Acceptability measured by self ratings of Acceptability of Intervention Measure (AIM)
Intervention Appropriateness | 1 month after implementation start
  Intervention Appropriateness measured by self ratings of Intervention Appropriateness Measure (IAM)
Intervention Appropriateness | 6 months after implementation start
  Intervention Appropriateness measured by self ratings of Intervention Appropriateness Measure (IAM)
Compliance to intervention | Summary of compliance 6 months after implementation start
  Compliance to intervention measured by weekly observations and reports of performed training activities
Normalization of intervention | 6 months after implementation start
  Normalization of intervention measured by The Swedish version of the Normalization Process Theory Measure (S-NoMAD)
Normalization of intervention | 1 year after implementation start
  Normalization of intervention measured by The Swedish version of the Normalization Process Theory Measure (S-NoMAD)
Normalization of intervention | 2 years after implementation start
  Normalization of intervention measured by The Swedish version of the Normalization Process Theory Measure (S-NoMAD)
Qualitative interviews | After the implementation phase i.e., 6 months after implementation start
  Qualitative interviews concerning acceptability, feasibility, appropriateness, compliance and normalization of the intervention

SECONDARY OUTCOMES:
Burnout | Change from baseline to follow up observation 6 months after inclusion
  Burnout measured by self ratings of Burnout Shirom-Melamed Burnout Questionnaire (SMBQ-6), scores 6-42, higher scores indicates more burnout symptoms
Burnout | Follow up 12 months after inclusion
  Burnout measured by self ratings of Burnout Shirom-Melamed Burnout Questionnaire (SMBQ-6), scores 6-42, higher scores indicates more burnout symptoms
Sleep difficulties | Change from baseline to follow up observation 6 months after inclusion
  Sleep difficulties measured by self ratings of Insomnia Severity Index (ISI), , scores 0-28, higher scores indicates more sleep difficulties
Sleep difficulties | Follow up 12 months after inclusion
  Sleep difficulties measured by self ratings of Insomnia Severity Index (ISI), , scores 0-28, higher scores indicates more sleep difficulties
Work and illness | Change from baseline to follow up observation 6 months after inclusion
  Work and illness measured by section C of Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P)
Work and illness | Follow up 12 months after inclusion
  Work and illness measured by section C of Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P)
Engagement at work | Change from baseline to follow up observation 6 months after inclusion
  Engagement at work measured by Utrecht work engagement scale (UWES-9S), scores 0-54, higher scores indicates more work engagement
Engagement at work | Follow up 12 months after inclusion
  Engagement at work measured by Utrecht work engagement scale (UWES-9S), scores 0-54, higher scores indicates more work engagement
Minutes spent on Physical movement (high, moderate, low) | Follow up observation 12 months after inclusion
  Physical exercise conducted by staff, measured by actigraph
Minutes spent on Physical movement (high, moderate, low) | Follow up 12 months after inclusion
  Physical exercise conducted by staff, measured by self ratings of International Physical Activity Questionnaires (IPAQ)
General health | Follow up 12 months after inclusion
  General health measured by self ratings of General health questionnaire (GHQ), scores 0-12, higher scores indicates more mental distress
Perceived stress | Follow up 12 months after inclusion
  Perceived stress measured by self ratings of Perceived stress scale (PSS-10), , scores 0-40, higher scores indicates more mental distress
Ratings of Braining sessions | During the period intervention start to 6 months follow up
  Self constructed questions where staff rate how many Braining sessions they have attended per week.
Ratings of Braining sessions | During the period 6 months follow up to 12 months follow up
  Self constructed questions where staff rate how many Braining sessions they have attended per week.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Martinsson, PhD, Principal Investigator — Region Stockholm and Karolinska institiutet
Locations (1):
- Region Stockholm, Liljeholmsberget, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No